CLINICAL TRIAL: NCT07249775
Title: AI-Driven Early Detection of Cachexia in Pancreatic Cancer and Feasibility of Diet and Exercise Interventions
Brief Title: A First-in-Human Study of FID-022 in Solid Tumor Patients
Status: Recruiting | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Florida Cancer Innovation Fund (Unknown)
Responsible Party: Sponsor
Other Study IDs: MCC-23812
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Cancer Cachexia
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic Cancer Patients: Patients with newly diagnosed borderline resectable or locally advanced pancreatic adenocarcinoma.
  Interventions: Other: Baseline Lifestyle and Symptom Assessment; Other: Extended Lifestyle Monitoring
- Oncology Clinicians: Medical oncologists, APPs, dietitians involved in pancreatic cancer care.
  Interventions: Other: Feasibility Survey

INTERVENTIONS:
Other: Baseline Lifestyle and Symptom Assessment — Dietary questionnaire (VioScreen), symptom and QoL surveys (ESAS-r, FAACT, PROMIS PF, PG-SGA), physical activity survey (Modified GLTEQ), functional fitness tests, DEXA scans, blood draws.
  Groups: Pancreatic Cancer Patients
Other: Extended Lifestyle Monitoring — Wearable monitoring (Fitbit) and diet/physical activity preference survey at 9 months.
  Groups: Pancreatic Cancer Patients
Other: Feasibility Survey — One-time structured survey assessing integration of diet and exercise interventions into clinical workflow.
  Groups: Oncology Clinicians

SUMMARY:
This observational study aims to (1) validate a multimodal artificial intelligence (AI) model for early detection of cancer-associated cachexia in pancreatic cancer patients and (2) assess the feasibility and acceptability of diet and exercise interventions for cachexia management. The study will use retrospective data from the Florida Pancreas Collaborative and prospective data from newly diagnosed patients at Moffitt Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically confirmed diagnosis of pancreatic exocrine malignancy (e.g.pancreatic ductal adenocarcinoma, acinar cell carcinoma, pancreatic adenosquamous carcinoma, etc.) or clinical features highly suggestive of such malignancy with diagnostic confirmation anticipated during the screening or early study period.
* Presentation consistent with resectable, borderline resectable, local, or locally advanced, or metastatic disease
* May or may not have had surgery
* Treatment plan likely includes systemic therapy for pancreatic cancer
* ECOG performance status 0-2
* Able to tolerate oral intake and not currently receiving enteral or parenteral nutrition
* Able to read and speak English
* Able to provide written informed consent

Exclusion Criteria:

* Pregnant or breastfeeding at the time of enrollment
* Current use of tube feeding (enteral) or total parenteral nutrition
* Presence of ascites or other findings suggestive of decompensated disease
* Evidence or history of bowel obstruction or any gastrointestinal condition that may limit food intake
* Severe or uncontrolled psychiatric illness (e.g., psychosis, dementia) that would interfere with participation
* Presence of other uncontrolled intercurrent illnesses (e.g., infection, heart failure, liver failure) that may interfere with protocol adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years) with histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC), presenting with resectable, borderline resectable, or locally advanced nonmetastatic disease. ECOG performance status 0-2. Total enrollment includes 100 newly diagnosed pancreatic cancer patients (cross-sectional), a longitudinal subset of 50 patients followed for 9 months, and 20 oncology clinicians completing feasibility surveys.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
AI Model Performance | Up to 9 months
  Investigators will rigorously assess model performance using clinically meaningful metrics (AUC-ROC, sensitivity, specificity, etc.) to confirm its reliability and readiness for clinical use.
Survey Completion Rate | Up to 9 months
  Percentage of patients completing all scheduled questionnaires.
Wearable Adherence | Up to 9 months
  Percentage of longitudinal participants syncing Fitbit weekly for ≥80% of study weeks.
Quality of Life Change | Up to 9 months
  Mean change in FAACT total score from baseline to 9 months.
Physical Activity Change | Up to 9 months
  Mean increase in weekly moderate-to-vigorous activity minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rasool, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States